CLINICAL TRIAL: NCT05224193
Title: Physical ACTIVity, slEep, Fitness and Quality of Life in Children and Adolescents With Inflammatory Bowel Disease: a 5-year Prospective Observational Cohort Study - The ACTIVE-IBD Study
Brief Title: ACTIVE-IBD Study: Physical Activity and Sleep in Paediatric Inflammatory Bowel Disease
Acronym: ACTIVE-IBD
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CHI1102; 301029 (Other: IRAS)
Record Dates: First submitted 2021-09-16; First posted 2022-02-04 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Inflammatory Bowel Diseases; Exercise
Keywords: Exercise; Sleep; Quality of Life; Physical Activity
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric Patients with Inflammatory Bowel Disease

SUMMARY:
Assessment of physical activity on children with Inflammatory Bowel Disease using questionnaires and wrist watch based activity monitors.

The participants will be recruited from paediatric IBD clinics and will undergo questionnaires to assess their activity level, disease activity and quality of life scores. The participants will then be invited to wear a wrist based accelerometer for a week. The participants will complete a physical activity diary, food diary and stool chart at the same time.

Results will be analysed to see the level of physical activity and assess if the participants are meeting the recommended level of physical activity

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents from age of 6 to 18 years of age
* Confirmed endoscopic/histology based IBD diagnosis
* Under the care of the Southampton University Hospitals NHS Foundation Trust paediatric gastroenterology team
* Able to provide consent / assent to participate in the study
* Able to understand and/or cooperate with the study requirements
* Pregnant participants will be included as long as they can complete the physical assessmentsExclusion Criteria:

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any disease known to interfere with exercise:
  * poorly controlled asthma
  * significant cardiovascular disease
  * fracture
  * infection
    * Unable to understand and/or cooperate with the study requirements
    * Unable to provide consent / assent to participate in the study
    * Participants will eb excluded if they are currently part of another exercise/ physical study
    * Unable to provide consent / assent to participate in study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Moderate Vigorous Physical Activity measurement | Over 1 Week
  Amount of time spent performing moderate and vigorous physical activity
Sedentary time | 1 week
  Amount of time spent sedentary

SECONDARY OUTCOMES:
Disease Activity | At Baseline Clinical Assessment
  Disease activity scores using either PUCAI (/85) or PCDAI (/100). Higher scores indicate more active disease
Perceived Physical Activity | At Baseline Clinical Assessment
  Youth Physical Activity Scale - Subjective Assessment of Moderate Vigorous Physical Activity in Hours over a 1 week retrospective period
Amount and Quality of Sleep | At Baseline Clinical Assessment
  Child Sleep Health Questionnaire scored out of 154 total and is parent/ carer subjective sleep assessment. Scored in four separate domains. Higher scores indicate increased duration and quality of sleep
Nutritional Assessment | At Baseline Clinical Assessment
  Mid Upper Arm Circumference
Growth Assessment | At Baseline Clinical Assessment
  Height in meters
Growth Assessment | At Baseline Clinical Assessment
  Weight in kg
Nutrition Assessment | 3 day assessment after baseline visit
  3 day self-reported food diary
Amount and Quality of Sleep | 1 week period
  Accelerometer measured sleep

OTHER OUTCOMES:
Quality of Life Score | At baseline clinic assessment
  Paediatric Quality of Life Score - PEDSQL scored in psychosocial and physical sections. Both are scored out of 100 and the higher the score the better health related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No